CLINICAL TRIAL: NCT03687723
Title: Observational Study of the Clinical Use of the Organ Care System (OCS™) in Heart Transplantation
Brief Title: Observational Study of the Clinical Use of the OCS™ Heart
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: OCS-Heart-2016
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: OCS Heart System — The OCS™ Heart System is a portable organ perfusion and monitoring medical device intended to preserve donor hearts in a near physiologic and beating state prior to transplantation.

SUMMARY:
Single-arm, prospective, multi-center observational study of the clinical use of the ex-vivo perfusion of the heart with the Organ Care System (OCS™)

DETAILED DESCRIPTION:
This is an observational study at two centers that will enroll minimum of 60 heart transplant recipients transplanted with donor heart preserved using the OCS™ Heart System. All consented subjects who receive OCS™-preserved heart transplants will be approached for participation. The study will evaluate short and long-term effectiveness of the OCS™ Heart System for heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

All recipients of heart transplantation with Use of the OCS™ Heart

Exclusion Criteria:

Donor Hearts

* Presence of coronary heart diseases
* acute myocardial infarction
* Presence of heart valve disease (Stenosis or Insufficiency > first degree)
* Presence of left ventricular hypertrophy (septum and posterior wall thickness >1.7 cm)
* State of shock of donor (MAP <60 mmHg, CVP >15, PCWP >15 mmHg) with use of Dobutamine >10 ug/kg/min and/or Norepinephrine > 0.5 ug/kg/min or Epinephrine > 0.2 ug/kg/min
* irreversible persistant pulmonary hypertrophy, defined as transpulmonary gradient >15 mmHg of the recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring heart transplantation who receive OCS™-preserved heart transplants.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Patient Survival | 12 months
  12-month patient survival post heart transplant Primary Effectiveness Endpoint

SECONDARY OUTCOMES:
Patient and Graft Survival | 30 days
  30-day patient and graft survival post heart transplant

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ius, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Department of Cardiothoracic, Transplant and Vascular Surgery, Hanover, Germany